CLINICAL TRIAL: NCT00868439
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Parallel-Group, Multiple-Dose Study to Evaluate the Effects of Patiromer in Heart Failure Patients
Brief Title: Evaluation of Patiromer in Heart Failure Patients
Acronym: PEARL-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Relypsa, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RLY5016-202
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hyperkalemia; Heart Failure
Keywords: HF; Heart failure; hyperkalemia; chronic kidney disease; prevention of hyperkalemia in heart failure participants
MeSH Terms: conditions — Hyperkalemia; Heart Failure; Renal Insufficiency, Chronic | interventions — patiromer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- patiromer (Active Comparator)
  Interventions: Drug: patiromer
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: patiromer — Active investigational drug
  Other Names: RLY5016; Veltassa
  Arms: patiromer
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study was to assess the effects of patiromer on serum potassium participants with heart failure. This study also assessed the safety and tolerability of patiromer in participants with heart failure.

DETAILED DESCRIPTION:
This was a double-blind, randomized, placebo-controlled, parallel-group, multiple-dose study in congestive heart failure participants. Depending on the outcome from the initial cohort of 100 participants (Part 1), a second cohort of 170 participants could have been enrolled (Part 2). Based on the results of Part 1 of the study, Part 2 was not conducted.

Participants were randomly assigned to and received patiromer (30 g/day) or placebo for up to 28 days. All participants also received spironolactone; the initial spironolactone dose was 25 mg daily and was increased to 50 mg daily for participants who had a serum potassium ≤ 5.1 mEq/L on treatment Day 14. Study visits occurred on treatment Days 3, 7, 14, 17, 21 and 28. A safety follow-up contact was made 7 days after administration of last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic heart failure clinically indicated to receive spironolactone therapy, aged 18 years or older with serum potassium level of 4.3 - 5.1 mEq/L at screening and baseline, AND (1) chronic kidney disease (GFR < 60 mL/min) OR (2) documented history of hyperkalemia within the last 6 months
* Females of child-bearing potential must be non-lactating, must have a negative serum pregnancy test at screening, and must have used a highly effective form of contraception for at least 3 months before study drug administration, during the study, and for one month after study completion
* Male participants and/or their female partners of child-bearing potential must use a highly effective form of contraception during the study and for 3 months after study completion
* Must sign informed consent document

Exclusion Criteria:

* History of bowel obstruction, swallowing disorders, severe gastrointestinal disorders or major gastrointestinal surgery
* Uncorrected hemodynamically significant primary valvular disease, known obstructive or restrictive cardiomyopathy, uncontrolled or hemodynamically unstable arrhythmia
* Coronary-artery bypass graft, percutaneous intervention (e.g. cardiac, cerebrovascular, aortic), or major surgery including thoracic and cardiac, within 3 months prior to baseline or anticipated need during study participation
* Heart transplant recipient, or anticipated need for transplant during study participation
* Any of the following events having occurred within 3 months prior to baseline: unstable angina as judged by the Investigator, unresolved acute coronary syndrome, transient ischemic attack or stroke
* Current dialysis participant, or anticipated need for dialysis during study participation
* Prior kidney transplant, or anticipated need for transplant during study participation
* Metastatic, late-stage or end-stage cancer with < 12 months life expectancy
* History of alcoholism or drug/chemical abuse within 1 year
* QTcB interval > 500 msec (Bazett's correction formula)
* Sustained systolic blood pressure > 170 or < 90 mmHg
* Liver enzymes (ALT, AST) > 3 times upper limit of normal
* Use of oral cardiac medications (including loop and thiazide diuretics) that have not been stable for at least 21 days prior to baseline and are not anticipated to remain stable during study participation
* Use of any IV cardiac medications within 21 days prior to baseline, or their anticipated need during study participation.
* Current use of polymer-based drugs (e.g. Renagel, Kayexalate, Welchol, Colestid), other phosphate binders or potassium binders, calcium supplements, antacids (eg TUMS, Maalox), or their anticipated need during study participation
* Use of aldosterone antagonist in the last 30 days prior to baseline, unless was discontinued due to hyperkalemia
* Use of potassium sparing medication and/or potassium supplements in the last 30 days prior to baseline
* Use of any investigational medication, 30 days or 5 half-lives whichever is longer, prior to baseline
* Participants who have taken investigational product in this study, or a previous patiromer study
* Inability to consume the study medication, or, in the opinion of the Investigator, inability to comply with the protocol
* In the opinion of the Investigator, any medical condition, uncontrolled systemic disease, serious intercurrent illness, or extenuating circumstance occurring or persisting, within 30 days prior to baseline, that would significantly decrease study compliance or jeopardize the safety of the participant or affect the validity of the trial results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Operations, Study Director — Relypsa, Inc.
Locations (33):
- United States (9):
  - Investigator Site 029, Miami, Florida
  - Investigator Site 031, Port Charlotte, Florida
  - Investigator Site 009, Peoria, Illinois
  - Investigator Site 018, Minneapolis, Minnesota
  - Investigator Site 020, Buffalo, New York
  - Investigator Site 005, Northport, New York
  - Investigator Site 022, Columbus, Ohio
  - Investigator Site 001, Dallas, Texas
  - Investigator Site 019, Salt Lake City, Utah
- Czechia (3):
  - Investigator Site 102, Brno
  - Investigator Site 104, Prague
  - Investigator Site 103, Prague
- Georgia (4):
  - Investigator Site 605, Tbilisi
  - Investigator Site 602, Tbilisi
  - Investigator Site 604, Tbilisi
  - Investigator Site 603, Tbilisi
- Germany (2):
  - Investigator Site 201, Göttingen
  - Investigator Site 202, Heidelberg
- Investigator Site 305, Warsaw, Poland
- Russia (8):
  - Investigator Site 409, Barnaul
  - Investigator Site 407, Kemerovo
  - Investigator Site 406, Moscow
  - Investigator Site 402, Moscow
  - Investigator Site 403, Moscow
  - Investigator Site 404, Saint Petersburg
  - Investigator Site 412, Saint Petersburg
  - Investigator Site 405, Saint Petersburg
- Ukraine (6):
  - Investigator Site 507, Dnipropetrovsk
  - Investigator Site 502, Kharkiv
  - Investigator Site 509, Kharkiv
  - Investigator Site 504, Kiev
  - Investigator Site 506, Kiev
  - Investigator Site 501, Kiev

REFERENCES:
- [Result] Pitt B, Anker SD, Bushinsky DA, Kitzman DW, Zannad F, Huang IZ; PEARL-HF Investigators. Evaluation of the efficacy and safety of RLY5016, a polymeric potassium binder, in a double-blind, placebo-controlled study in patients with chronic heart failure (the PEARL-HF) trial. Eur Heart J. 2011 Apr;32(7):820-8. doi: 10.1093/eurheartj/ehq502. Epub 2011 Jan 5. PMID 21208974
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 subjects were randomized in Part 1 of the study (60 to each treatment group). Of these, 120 randomized subjects, 105 received either RLY5016 Powder for Suspension (n = 56) or placebo (n = 49).
Pre-assignment Details: Eligible participants ≥ 18 y/o, had history of chronic HF, clinically initiated spironolactone therapy, serum K+ = 4.3 - 5.1 mEq/L at screening and baseline, and either had 1) CKD, w/ eGFR < 60 mL/min and receiving HF therapies or 2) documented history of hyperkalemia led to discontinuation w/ aldosterone antagonist w/in 6 months prior to baseline.
Groups:
- Patiromer: Spironolactone + Patiromer
  Participants received patiromer (15 g twice daily [BID]).
  Participants also started spironolactone at a dose of 25 mg/day, which was increased to 50 mg/day after 2 weeks if the participant's serum potassium (based on local laboratory determination) was > 3.5 mEq/L and ≤ 5.1 mEq/L. The spironolactone dose remained at 25 mg/day if the serum potassium was > 5.1 mEq/L and ≤ 5.5 mEq/L. If, at any time, a participant's serum potassium level was confirmed to be ≤ 3.5 mEq/L or > 5.5 mEq/L based on local laboratory data, the participant was to be discontinued from the study.
- Placebo: Spironolactone + Placebo
  Participants received placebo (twice daily [BID]).
  Participants also started spironolactone at a dose of 25 mg/day, which was increased to 50 mg/day after 2 weeks if the participant's serum potassium (based on local laboratory determination) was > 3.5 mEq/L and ≤ 5.1 mEq/L. The spironolactone dose remained at 25 mg/day if the serum potassium was > 5.1 mEq/L and ≤ 5.5 mEq/L. If, at any time, a participant's serum potassium level was confirmed to be ≤ 3.5 mEq/L or > 5.5 mEq/L based on local laboratory data, the participant was to be discontinued from the study.
Period: Overall Study
Arm/Group | Patiromer | Placebo
Started | 56 | 49
Completed | 48 | 40
Not Completed | 8 | 9
Not completed — Adverse Event | 4 | 3
Not completed — Prot-Specified W/D Criteria (Serum K+) | 2 | 3
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant received one dose of patiromer and did not return to the clinic in a timely manner; the participant was terminated from the study for protocol noncompliance, and because the participant did not have post-treatment efficacy data, the participant was excluded from the Full Analysis Set but retained in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patiromer | Placebo | Total
Number analyzed (Participants) | 55 | 49 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 39 | 35 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (8.66) | 68.2 (10.46) | 68.3 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 15 | 41
  Male | 29 | 34 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Potassium to the End of the 28-day Treatment Period.
Time Frame: Baseline and Day 28
Population: Analysis was determined using Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 55 | 49
mEq/L | -0.21 (0.066) | 0.23 (0.072)
Statistical Analysis 1: Comparison: Patiromer vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Proportion of Participants With a Serum Potassium Level During the 28-day Treatment Period That Was > 5.5 mEq/L.
Description: Analysis based on central laboratory data.
Time Frame: 28 Days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 55 | 49
percentage of participants | 7.3 | 24.5
Statistical Analysis 1: Comparison: Patiromer vs Placebo; Test type: Superiority or Other; p = 0.027, Fisher Exact

3. Secondary Outcome: Proportion of Participants Discontinuing the Study Due to Serum Potassium Elevation (Serum K+ > 5.5 mEq/L).
Description: Analysis based on local laboratory data.
Time Frame: 28 Days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 55 | 49
percentage of participants | 0 | 6.1
Statistical Analysis 1: Comparison: Patiromer vs Placebo; Test type: Superiority or Other; p = 0.101, Fisher Exact

4. Secondary Outcome: Proportion of Participants Whose Spironolactone Dose Was Increased.
Time Frame: 28 Days
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 55 | 49
percentage of participants | 90.9 | 73.5
Statistical Analysis 1: Comparison: Patiromer vs Placebo; Test type: Superiority or Other; p = 0.022, Fisher Exact

5. Secondary Outcome: Proportion of Participants With an Increase in Serum Potassium Level From Baseline to the End of the 28-day Treatment Period That Was ≥ 0.5 mEq/L
Time Frame: Baseline and Day 28
Population: Analysis was determined using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 55 | 49
percentage of participants | 12.7 | 24.5
Statistical Analysis 1: Comparison: Patiromer vs Placebo; Test type: Superiority or Other; p = 0.136, Fisher Exact

6. Secondary Outcome: Time to First Elevated Serum K+ > 5.5 mEq/L.
Time Frame: 28 Days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 55 | 49
days | NA [NA to NA] — Median time for first occurrence of serum potassium > 5.5 mEq/L was not reached. | NA [NA to NA] — Median time for first occurrence of serum potassium > 5.5 mEq/L was not reached.
Statistical Analysis 1: Comparison: Patiromer vs Placebo; Test type: Superiority or Other; p = 0.015, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 7 days after Day 28 or last patiromer dose, whichever was earlier.
Description: Randomized participants who received at least one dose of trial medication.
Arm/Group | Patiromer | Placebo
Serious Adverse Events (participants affected / at risk) | 2/56 | 2/49
Other Adverse Events (participants affected / at risk) | 11/56 | 1/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer (N=56) | Placebo (N=49)
Coronary artery disease (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer (N=56) | Placebo (N=49)
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 4 | 0
Blood urea increased (Investigations) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements generally provide that PI cannot publish single site data before publication of the multi-site publication, unless 1 year has elapsed since completion of the study at all sites. Thereafter, PI may publish provided that PI shall: provide a copy of the publication to sponsor at least 60 days in advance of submission for publication; delete sponsor's confidential information as requested; and delay publication up to an additional 90 days to permit protection of intellectual property.